CLINICAL TRIAL: NCT03234842
Title: A Phase II Trial of Dose Escalated Proton Beam Therapy or Photon Therapy for Resectable and Unresectable Esophageal Cancer
Brief Title: Dose Escalated Proton Beam Therapy or Photon Therapy for Esophageal Cancer
Acronym: ES01
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: non-accrual
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 1605-ES01
Record Dates: First submitted 2017-07-21; First posted 2017-07-31 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Esophageal Cancer
Keywords: Esophagus; Proton; Radiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Proton Therapy; Drug Therapy; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Proton (Experimental): Proton beam therapy of 59.4 Gy in 1.8 Gy fractions (50.4 Gy if unable to meet cardiac/lung- organs at risk (OAR) constraints) plus concurrent standard chemotherapy
  Interventions: Radiation: Proton Beam Therapy; Drug: Chemotherapy
- Photon (Active Comparator): Photon Radiation therapy of 59.4 Gy in 1.8Gy fractions ( 50.4 Gy if unable to meet cardiac/lung- organs at risk (OAR) constraints) plus concurrent standard chemotherapy
  Interventions: Radiation: Photon Radiation Therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — 59.4 Gy (RBE) in 1.8 Gy per fraction plus weekly chemotherapy at standard doses
  Other Names: Proton Therapy
  Arms: Proton
Radiation: Photon Radiation Therapy — 59.4 Gy (RBE) in 1.8 Gy per fraction plus weekly chemotherapy at standard doses
  Other Names: IMRT
  Arms: Photon
Drug: Chemotherapy — Concurrent weekly chemotherapy at standard doses
  Other Names: Carboplatin; Paclitaxel

SUMMARY:
This study will evaluate if proton beam therapy as part of chemoradiation results in a decrease in diffusion lung capacity of carbon monoxide (DLCO) compared to photon radiation therapy for esophageal carcinoma. A secondary objective is to determine effects on cardiac function, quality of life, and compare acute and late toxicities.

DETAILED DESCRIPTION:
Radiation Modality: Proton radiotherapy will be offered to all patients that meet trial eligibility. If patients decline proton radiotherapy or are otherwise unable to receive proton therapy they will be included in x-ray cohort (group 2).

Chemotherapy will be delivered at the discretion of the treating Medical Oncologist. Weekly carboplatin and paclitaxel at standard doses is preferred. It is recommended that the weekly chemotherapy regimen be continued throughout the course of radiotherapy. Chemotherapy should begin within 48 hours of beginning radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years at the time of consent.
* Pathologically confirmed esophageal adenocarcinoma or squamous cell. carcinoma of the thoracic esophagus or esophagogastric junction.
* Patient's preliminary cancer stage, according to the AJCC 7th edition staging, must be cT1b-T4, N0-N3.

Exclusion Criteria:

* Patients with cervical esophageal carcinoma.
* Prior radiotherapy with fields overlapping the current esophageal cancer.
* Patients with cT1a disease.
* Patients with evidence of tracheoesophageal fistula must undergo bronchoscopy to exclude fistula.
* Patients with distant metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Compare the rate of a clinically significant reduction of DLCO (defined as a decrease of ≥ 10% from baseline) between protons and photons after preoperative or definitive chemoradiation | Approximately 12 months after radiation therapy
  Participants with a clinically significant reduction of DLCO approximately 12 months after radiation therapy

SECONDARY OUTCOMES:
Compare quality of life | Approximately 12 months after radiation therapy
  Participants quality of life results using EORTC Quality of Life Questionnaire - Oesophageal Cancer Module (OES-18) and EORTC QLQ C-30 conjointly approximately 12 months after radiation therapy
Compare outcomes for local control | Approximately 12 months after radiation therapy
  Number of participants with local control for proton and photon radiation and concurrent chemotherapy as part of definitive therapy or trimodality therapy approximately 12 months after radiation therapy
Compare outcomes for progression free survival | Approximately 12 months after radiation therapy
  Number of participants with progression free survival for proton and photon radiation and concurrent chemotherapy as part of definitive therapy or trimodality therapy approximately 12 months after radiation therapy
Compare overall survival rates | Approximately 12 months after radiation therapy
  Number of participants with overall survival rates for proton and photon radiation and concurrent chemotherapy as part of definitive therapy or trimodality therapy approximately 12 months after radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rutenberg, MD, PhD, Principal Investigator — UF Health Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Walsh TN, Noonan N, Hollywood D, Kelly A, Keeling N, Hennessy TP. A comparison of multimodal therapy and surgery for esophageal adenocarcinoma. N Engl J Med. 1996 Aug 15;335(7):462-7. doi: 10.1056/NEJM199608153350702. PMID 8672151
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Background] Stahl M, Stuschke M, Lehmann N, Meyer HJ, Walz MK, Seeber S, Klump B, Budach W, Teichmann R, Schmitt M, Schmitt G, Franke C, Wilke H. Chemoradiation with and without surgery in patients with locally advanced squamous cell carcinoma of the esophagus. J Clin Oncol. 2005 Apr 1;23(10):2310-7. doi: 10.1200/JCO.2005.00.034. PMID 15800321
- [Background] Bedenne L, Michel P, Bouche O, Milan C, Mariette C, Conroy T, Pezet D, Roullet B, Seitz JF, Herr JP, Paillot B, Arveux P, Bonnetain F, Binquet C. Chemoradiation followed by surgery compared with chemoradiation alone in squamous cancer of the esophagus: FFCD 9102. J Clin Oncol. 2007 Apr 1;25(10):1160-8. doi: 10.1200/JCO.2005.04.7118. PMID 17401004
- [Background] Gergel TJ, Leichman L, Nava HR, Blumenson LE, Loewen GM, Gibbs JE, Khushalani NI, Leichman CG, Bodnar LM, Douglass HO, Smith JL, Kuettel MR, Proulx GM. Effect of concurrent radiation therapy and chemotherapy on pulmonary function in patients with esophageal cancer: dose-volume histogram analysis. Cancer J. 2002 Nov-Dec;8(6):451-60. doi: 10.1097/00130404-200211000-00009. PMID 12500854
- [Background] von Dobeln GA, Nilsson M, Adell G, Johnsen G, Hatlevoll I, Tsai J, Lundell L, Lund M, Lind P. Pulmonary function and cardiac stress test after multimodality treatment of esophageal cancer. Pract Radiat Oncol. 2016 May-Jun;6(3):e53-e59. doi: 10.1016/j.prro.2015.10.015. Epub 2015 Nov 10. PMID 26725962
- [Background] Lee HK, Vaporciyan AA, Cox JD, Tucker SL, Putnam JB Jr, Ajani JA, Liao Z, Swisher SG, Roth JA, Smythe WR, Walsh GL, Mohan R, Liu HH, Mooring D, Komaki R. Postoperative pulmonary complications after preoperative chemoradiation for esophageal carcinoma: correlation with pulmonary dose-volume histogram parameters. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1317-22. doi: 10.1016/s0360-3016(03)01373-7. PMID 14630268
- [Background] Wang J, Wei C, Tucker SL, Myles B, Palmer M, Hofstetter WL, Swisher SG, Ajani JA, Cox JD, Komaki R, Liao Z, Lin SH. Predictors of postoperative complications after trimodality therapy for esophageal cancer. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):885-91. doi: 10.1016/j.ijrobp.2013.04.006. PMID 23845841
- [Background] Lund M, Alexandersson von Dobeln G, Nilsson M, Winter R, Lundell L, Tsai JA, Kalman S. Effects on heart function of neoadjuvant chemotherapy and chemoradiotherapy in patients with cancer in the esophagus or gastroesophageal junction - a prospective cohort pilot study within a randomized clinical trial. Radiat Oncol. 2015 Jan 13;10:16. doi: 10.1186/s13014-014-0310-7. PMID 25582305
- [Background] De Jaeger K, Seppenwoolde Y, Boersma LJ, Muller SH, Baas P, Belderbos JS, Lebesque JV. Pulmonary function following high-dose radiotherapy of non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2003 Apr 1;55(5):1331-40. doi: 10.1016/s0360-3016(02)04389-4. PMID 12654445
- [Background] Marks LB, Fan M, Clough R, Munley M, Bentel G, Coleman RE, Jaszczak R, Hollis D, Anscher M. Radiation-induced pulmonary injury: symptomatic versus subclinical endpoints. Int J Radiat Biol. 2000 Apr;76(4):469-75. doi: 10.1080/095530000138466. PMID 10815626
- [Background] Lopez Guerra JL, Gomez DR, Zhuang Y, Levy LB, Eapen G, Liu H, Mohan R, Komaki R, Cox JD, Liao Z. Changes in pulmonary function after three-dimensional conformal radiotherapy, intensity-modulated radiotherapy, or proton beam therapy for non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):e537-43. doi: 10.1016/j.ijrobp.2012.01.019. Epub 2012 Mar 13. PMID 22420964
- [Background] Miller KL, Zhou SM, Barrier RC Jr, Shafman T, Folz RJ, Clough RW, Marks LB. Long-term changes in pulmonary function tests after definitive radiotherapy for lung cancer. Int J Radiat Oncol Biol Phys. 2003 Jul 1;56(3):611-5. doi: 10.1016/s0360-3016(03)00182-2. PMID 12788165
- [Background] Enache I, Noel G, Jeung MY, Meyer N, Oswald-Mammosser M, Pistea C, Jung GM, Mennecier B, Quoix E, Charloux A. Impact of 3D conformal radiotherapy on lung function of patients with lung cancer: a prospective study. Respiration. 2013;86(2):100-8. doi: 10.1159/000342371. Epub 2012 Nov 13. PMID 23154264
- [Background] Borst GR, De Jaeger K, Belderbos JS, Burgers SA, Lebesque JV. Pulmonary function changes after radiotherapy in non-small-cell lung cancer patients with long-term disease-free survival. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):639-44. doi: 10.1016/j.ijrobp.2004.11.029. PMID 15936539
- [Background] Ferguson MK, Celauro AD, Prachand V. Prediction of major pulmonary complications after esophagectomy. Ann Thorac Surg. 2011 May;91(5):1494-1500; discussion 1500-1. doi: 10.1016/j.athoracsur.2010.12.036. PMID 21524462
- [Background] Ferguson MK, Durkin AE. Preoperative prediction of the risk of pulmonary complications after esophagectomy for cancer. J Thorac Cardiovasc Surg. 2002 Apr;123(4):661-9. doi: 10.1067/mtc.2002.120350. PMID 11986593
- [Background] Lin FC, Durkin AE, Ferguson MK. Induction therapy does not increase surgical morbidity after esophagectomy for cancer. Ann Thorac Surg. 2004 Nov;78(5):1783-9. doi: 10.1016/j.athoracsur.2004.04.081. PMID 15511475
- [Background] Cerfolio RJ, Talati A, Bryant AS. Changes in pulmonary function tests after neoadjuvant therapy predict postoperative complications. Ann Thorac Surg. 2009 Sep;88(3):930-5; discussion 935-6. doi: 10.1016/j.athoracsur.2009.06.013. PMID 19699923
- [Background] Gill PG, Denham JW, Jamieson GG, Devitt PG, Yeoh E, Olweny C. Patterns of treatment failure and prognostic factors associated with the treatment of esophageal carcinoma with chemotherapy and radiotherapy either as sole treatment or followed by surgery. J Clin Oncol. 1992 Jul;10(7):1037-43. doi: 10.1200/JCO.1992.10.7.1037. PMID 1607911
- [Background] Chirieac LR, Swisher SG, Ajani JA, Komaki RR, Correa AM, Morris JS, Roth JA, Rashid A, Hamilton SR, Wu TT. Posttherapy pathologic stage predicts survival in patients with esophageal carcinoma receiving preoperative chemoradiation. Cancer. 2005 Apr 1;103(7):1347-55. doi: 10.1002/cncr.20916. PMID 15719440
- [Background] Meredith KL, Weber JM, Turaga KK, Siegel EM, McLoughlin J, Hoffe S, Marcovalerio M, Shah N, Kelley S, Karl R. Pathologic response after neoadjuvant therapy is the major determinant of survival in patients with esophageal cancer. Ann Surg Oncol. 2010 Apr;17(4):1159-67. doi: 10.1245/s10434-009-0862-1. Epub 2010 Feb 6. PMID 20140529
- [Background] Donahue JM, Nichols FC, Li Z, Schomas DA, Allen MS, Cassivi SD, Jatoi A, Miller RC, Wigle DA, Shen KR, Deschamps C. Complete pathologic response after neoadjuvant chemoradiotherapy for esophageal cancer is associated with enhanced survival. Ann Thorac Surg. 2009 Feb;87(2):392-8; discussion 398-9. doi: 10.1016/j.athoracsur.2008.11.001. PMID 19161745
- [Background] Bosset JF, Gignoux M, Triboulet JP, Tiret E, Mantion G, Elias D, Lozach P, Ollier JC, Pavy JJ, Mercier M, Sahmoud T. Chemoradiotherapy followed by surgery compared with surgery alone in squamous-cell cancer of the esophagus. N Engl J Med. 1997 Jul 17;337(3):161-7. doi: 10.1056/NEJM199707173370304. PMID 9219702
- [Background] Yoon DH, Jang G, Kim JH, Kim YH, Kim JY, Kim HR, Jung HY, Lee GH, Song HY, Cho KJ, Ryu JS, Kim SB. Randomized phase 2 trial of S1 and oxaliplatin-based chemoradiotherapy with or without induction chemotherapy for esophageal cancer. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):489-96. doi: 10.1016/j.ijrobp.2014.11.019. Epub 2015 Jan 30. PMID 25680595
- [Background] Spigel DR, Greco FA, Meluch AA, Lane CM, Farley C, Gray JR, Clark BL, Burris HA 3rd, Hainsworth JD. Phase I/II trial of preoperative oxaliplatin, docetaxel, and capecitabine with concurrent radiation therapy in localized carcinoma of the esophagus or gastroesophageal junction. J Clin Oncol. 2010 May 1;28(13):2213-9. doi: 10.1200/JCO.2009.24.8773. Epub 2010 Mar 29. PMID 20351330
- [Background] Ajani JA, Xiao L, Roth JA, Hofstetter WL, Walsh G, Komaki R, Liao Z, Rice DC, Vaporciyan AA, Maru DM, Lee JH, Bhutani MS, Eid A, Yao JC, Phan AP, Halpin A, Suzuki A, Taketa T, Thall PF, Swisher SG. A phase II randomized trial of induction chemotherapy versus no induction chemotherapy followed by preoperative chemoradiation in patients with esophageal cancer. Ann Oncol. 2013 Nov;24(11):2844-9. doi: 10.1093/annonc/mdt339. Epub 2013 Aug 23. PMID 23975663
- [Background] Venkat P, Shridhar R, Naghavi A, et al. Pathologic Complete Response and Dose Escalation with Preoperative Dose Painting IMRT Chemoradiation in Esophageal Cancer. IJROBP. 2015; 93:S219-220
- [Background] Makishima H, Ishikawa H, Terunuma T, Hashimoto T, Yamanashi K, Sekiguchi T, Mizumoto M, Okumura T, Sakae T, Sakurai H. Comparison of adverse effects of proton and X-ray chemoradiotherapy for esophageal cancer using an adaptive dose-volume histogram analysis. J Radiat Res. 2015 May;56(3):568-76. doi: 10.1093/jrr/rrv001. Epub 2015 Mar 9. PMID 25755255
- [Background] Wang J, Palmer M, Bilton SD, et al. Comparing Proton Beam to Intensity Modulated Radiation Therapy Planning in Esophageal Cancer. Int J Particle Ther. 2015;1:866-877.
- [Background] Wang SL, Liao Z, Vaporciyan AA, Tucker SL, Liu H, Wei X, Swisher S, Ajani JA, Cox JD, Komaki R. Investigation of clinical and dosimetric factors associated with postoperative pulmonary complications in esophageal cancer patients treated with concurrent chemoradiotherapy followed by surgery. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):692-9. doi: 10.1016/j.ijrobp.2005.08.002. Epub 2005 Oct 19. PMID 16242257
- [Background] Wei X, Liu HH, Tucker SL, Wang S, Mohan R, Cox JD, Komaki R, Liao Z. Risk factors for pericardial effusion in inoperable esophageal cancer patients treated with definitive chemoradiation therapy. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):707-14. doi: 10.1016/j.ijrobp.2007.10.056. Epub 2008 Jan 11. PMID 18191334
- [Background] Donohoe CL, McGillycuddy E, Reynolds JV. Long-term health-related quality of life for disease-free esophageal cancer patients. World J Surg. 2011 Aug;35(8):1853-60. doi: 10.1007/s00268-011-1123-6. PMID 21553202
- [Background] Blazeby JM, Conroy T, Hammerlid E, Fayers P, Sezer O, Koller M, Arraras J, Bottomley A, Vickery CW, Etienne PL, Alderson D; European Organisation for Research and Treatement of Cancer Gastrointestinal and Quality of Life Groups. Clinical and psychometric validation of an EORTC questionnaire module, the EORTC QLQ-OES18, to assess quality of life in patients with oesophageal cancer. Eur J Cancer. 2003 Jul;39(10):1384-94. doi: 10.1016/s0959-8049(03)00270-3. PMID 12826041
- [Background] Derogar M, Lagergren P. Health-related quality of life among 5-year survivors of esophageal cancer surgery: a prospective population-based study. J Clin Oncol. 2012 Feb 1;30(4):413-8. doi: 10.1200/JCO.2011.38.9791. Epub 2012 Jan 3. PMID 22215745
- [Background] Hurmuzlu M, Aarstad HJ, Aarstad AK, Hjermstad MJ, Viste A. Health-related quality of life in long-term survivors after high-dose chemoradiotherapy followed by surgery in esophageal cancer. Dis Esophagus. 2011 Jan;24(1):39-47. doi: 10.1111/j.1442-2050.2010.01104.x. Epub 2010 Sep 2. PMID 20819100
- [Background] Kachnic LA, Winter K, Wasserman T, Kelsen D, Ginsberg R, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Willett CG, Minsky BD. Longitudinal Quality-of-Life Analysis of RTOG 94-05 (Int 0123):A Phase III Trial of Definitive Chemoradiotherapy for Esophageal Cancer. Gastrointest Cancer Res. 2011 Mar;4(2):45-52. PMID 21673875
- [Background] Warren S, Partridge M, Carrington R, Hurt C, Crosby T, Hawkins MA. Radiobiological determination of dose escalation and normal tissue toxicity in definitive chemoradiation therapy for esophageal cancer. Int J Radiat Oncol Biol Phys. 2014 Oct 1;90(2):423-9. doi: 10.1016/j.ijrobp.2014.06.028. PMID 25304796